CLINICAL TRIAL: NCT05302622
Title: Determination of the Most Efficacious Period for the Use of Laparoscopic Simulators in Obstetrics and Gynecology Specialty Training
Brief Title: Detecting the Most Efficient Residency Time for Laparoscopic Simulators
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ahkam Göksel Kanmaz, Associated Professor, Tepecik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021/10-48
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Laparoscopy; Simulation Training

STUDY DESIGN:
Intervention Model Description: There is three group based on the surgical skills and ob/gyn residency years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Other): Have surgical experience both laparoscopy and laparotomy and senior resident
  Interventions: Other: There is no intervention planning
- Group 2 (Other): Have surgical skills only laparotomic gynecologic procedures and in the middle of his/her residency
  Interventions: Other: There is no intervention planning
- Group 3 (Other): Have no surgical experience on gynecologic procedures and newbie residents
  Interventions: Other: There is no intervention planning

INTERVENTIONS:
Other: There is no intervention planning — There is no intervention planning

SUMMARY:
Laparoscopic surgeries is one of the most common surgery in gynecologic procedures. Nowadays there are many laparoscopic simulators for training residents. In this study it is aimed to determine the most efficient residency year for laparoscopic simulators.

This study planned as a prospective study. There will be three group which include ob/gyn residents. The residents will choose based on their residency year and surgery skills. 1. The residents who makes surgeries both laparoscopic and laparotomic, 2. The residents who makes surgeries only laparotomic, 3. The residents who won't any gynecologic surgery The data of surgery time, complications and movement numbers will take from the simulator. Tubal ligation and salpingooferectomy choose for the surgery examples. The simulation results of participants will compare and try to find the best improvement term for residency.

ELIGIBILITY:
Inclusion Criteria:

* Should be an ob/gyn resident
* Should except to participate study

Exclusion Criteria:

* Not to complete all simulations

Ages: 24 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Laparoscopic surgical procedures time | 6 months

SECONDARY OUTCOMES:
Movement number for laparoscopic procedures | 6 months
Complication during laparoscopic surgery simulations | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Education and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No